CLINICAL TRIAL: NCT03729570
Title: Testing an Electronic Pre-exposure Prophylaxis (PrEP) Initiation and Maintenance Home Care System to Promote PrEP Among Adolescent Men Who Have Sex With Men (MSM) in Rural and Small Town Areas
Brief Title: Electronic Pre-exposure Prophylaxis (PrEP) Initiation and Maintenance Home Care System
Acronym: ePrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of North Carolina, Chapel Hill (Other); University of Mississippi Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Aaron Siegler, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00103988; 3U19HD089881 (NIH)
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pre-exposure Prophylaxis
Keywords: PrEP; MSM; HIV; telemedicine; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ePrEP (Experimental): Participants will receive the ePrEP home care system for telemedicine PrEP, permitting initiation and persistence in PrEP care. The ePrEP home care system consists of: a smartphone application (app) for video-based telemedicine PrEP consultations with a clinician; secure messaging; a system to track shipments to & from participants; and behavioral risk surveys that are complemented by home specimen kits. Self-collected specimens will be mailed to laboratories for routine, guideline-based testing for PrEP care. Home specimen collection will be used to determine the primary study outcome of tenofovir-diphosphate levels.
  Interventions: Other: ePrEP
- Standard of care (No Intervention): Participants will be referred to a publicly available website that geolocates the nearest PrEP provider. They will receive standard of care, defined as what a member of the general public would be able to access for PrEP services. Home specimen self-collection will be used to determine the primary study outcome of tenofovir-diphosphate levels. Additional research assessments will include quarterly surveys.

INTERVENTIONS:
Other: ePrEP — Participants will have a baseline teleconsultation with a site study clinician who will be responsible for prescribing PrEP as indicated. They will be offered a 1-month check-in and telemedicine consultations at 3, 6, 9 and 12 months. Participants will complete home specimen collection for laboratory tests for each consultation. The virtual study visit consists of surveys, specimen collection, and a telemedicine consultation.
  Arms: ePrEP

SUMMARY:
The premise for the study is that a tailored approach for rural young men who have sex with men (YMSM), addressing known barriers of transportation, access to providers, and privacy, is most likely to yield high levels of Pre-exposure Prophylaxis (PrEP) initiation and persistence in care.

DETAILED DESCRIPTION:
The premise for the study is that a tailored approach for YMSM from rural and small town areas, addressing known barriers of transportation, access to providers, and privacy, is most likely to yield high levels of PrEP initiation and persistence in care. The study sites are Alabama, Georgia, North Carolina, and Mississippi.

Using a smartphone application (app), participants assigned to the intervention will receive and maintain a PrEP prescription without needing to leave their home (excepting pharmacy pick-up in some cases) - achieved through app-based surveys/screenings, telemedicine consultations, and home specimen self-collection.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male at birth
* Age 18-29 (inclusive)
* Live in a study state (Georgia, Mississippi, North Carolina, Alabama)
* Able to provide informed consent and complete survey instruments in English
* Willing to provide complete contact information (including 2 alternate contacts)
* Able and willing to provide identification verification for viewing confirmation only
* Laboratory confirmed HIV negative
* Owns a smartphone capable of running the study app
* Male sex partners in past 6 months or clinician discretion of epidemiologic context of HIV risk
* Behavioral/epidemiological indication for PrEP :

  * History of inconsistent or no condom use with more than one partner
  * History of inconsistent or no condom use with one partner who is not mutually monogamous
  * HIV-positive sexual partner
  * Any sexually transmitted infection (STI) diagnosed in past 6 months
  * Commercial sex work
  * African American MSM reporting anal sex in the past 6 months
  * Clinician discretion based on epidemiologic context of HIV risk
* Willing to take FDA-approved daily oral PrEP
* Willing to use study-provided PrEP navigation services
* Willing to self-collect specimens

Exclusion Criteria:

* HIV positive (self-report or laboratory confirmed)
* Chronic Hepatitis B or no verification of hepatitis B vaccination
* Currently enrolled in any HIV prevention trial (biomedical)
* Currently taking oral PrEP based on self-report
* Creatinine clearance <60 ml/min based on the Cockcroft-Gault equation
* Symptoms of acute HIV infection within the prior 30 days
* Contraindications to oral PrEP
* Personal diagnosis or family history of hemophilia
* Health insurance with Kaiser Permanente (unable to prescribe PrEP through the study)
* Investigator discretion to exclude anyone whose best interest is not to participate
* Evidence of fraudulent participation, such as duplicate Internet Protocol (IP) address, multiple screening attempts, duplicate emails, etc

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 217 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Siegler, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rollins School of Public Health, Atlanta, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Siegler AJ, Brock JB, Hurt CB, Ahlschlager L, Dominguez K, Kelley CF, Jenness SM, Wilde G, Jameson SB, Bailey-Herring G, Mena LA. An Electronic Pre-Exposure Prophylaxis Initiation and Maintenance Home Care System for Nonurban Young Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jun 10;8(6):e13982. doi: 10.2196/13982. PMID 31199326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited online in Georgia, North Carolina, Alabama, and Mississippi. Participating universities: Rollins School of Public Health in Atlanta, Georgia; University of North Carolina in Chapel Hill, North Carolina; University of Alabama in Birmingham, Alabama; and University of Mississippi Medical Center in Jackson, Mississippi. Enrollment began on May 28, 2019, and follow-up was complete by May 31, 2022. Study completion is defined as enrolled persons completing their 6-month survey.
Period: Overall Study
Arm/Group | ePrEP | Standard of Care
Started | 108 | 109
Completed | 80 | 84
Not Completed | 28 | 25
Not completed — Lost to Follow-up | 16 | 20
Not completed — Seroconversion | 5 | 0
Not completed — Moved out of the city | 1 | 0
Not completed — Time Conflict | 1 | 0
Not completed — Time Commitment | 2 | 0
Not completed — Bad Experience | 0 | 1
Not completed — No reason provided | 2 | 1
Not completed — Family Conflict | 0 | 1
Not completed — Did not want to continue taking medications | 0 | 1
Not completed — Found another PrEP provider | 1 | 0
Not completed — Did not enjoy being in the control group | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ePrEP | Standard of Care | Total
Number analyzed (Participants) | 108 | 109 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.29 (3.11) | 23.49 (3.24) | 23.39 (3.17)
Age, Customized [Count of Participants; unit: Participants]
  18 to 21 YO | 36 | 34 | 70
  22 to 25 YO | 42 | 43 | 85
  26 to 29 YO | 30 | 32 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 108 | 109 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 20
  Not Hispanic or Latino | 100 | 97 | 197
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 1 | 3 | 4
  Black or African American | 46 | 49 | 95
  White | 50 | 49 | 99
  Native American/Alaska Native | 1 | 1 | 2
  More than one race | 10 | 7 | 17
  Unknown or not reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 109 | 217

OUTCOME MEASURES:

1. Primary Outcome: Difference in Tenofovir-diphosphate (TFV-DP) Levels Between Intervention and Control Arms at 6 Months Follow-up
Description: Measurements TFV-DP levels will be conducted for participants in both arms using liquid chromatography/tandem mass spectrometry methods on self-collected DBS samples. TFV-DP level can be translated to an interpretation that indicates the mean number of days per week PrEP is ingested over approximately 1 month preceding specimen collection. The cutpoint used for the primary outcome measure will be medication levels indicating >4 doses/wk. For participants taking emtricitabine/tenofovir disoproxil fumarate, this will be TFV-DP levels: >1000 femtomole per blood spot (fmol/punch). For participants taking emtricitabine/tenofovir alafenamide this will be TFV-DP levels: >140 femtomole per blood spot (fmol/punch).
Time Frame: 6-month follow up
Population: Participants with biomarker data indicating adherent daily PrEP dosing. For participants either reporting the use of both medications in the period or not reporting which medication they used during this period, investigators used decision rules to determine adherence. For instance, if a participant had a TFV-DP level above both cutpoints, they were classified as adherent.
Measure: Count of Participants; unit: Participants
Arm/Group | ePrEP | Standard of Care
Number analyzed (Participants) | 31 | 26
Participants | 17 | 7

2. Secondary Outcome: Difference in Tenofovir-diphosphate (TFV-DP) Levels Between Intervention and Control Arms at 12 Months Follow-up
Description: Measurement of TFV-DP levels will be conducted for participants in both arms using liquid chromatography/tandem mass spectrometry methods on self-collected DBS samples. TFV-DP level can be translated to an interpretation that indicates the mean number of days per week PrEP is ingested over approximately 1 month preceding specimen collection. The cutpoint used for the primary outcome measure will be medication levels indicating >4 doses/wk. For participants taking emtricitabine/tenofovir disoproxil fumarate, this will be TFV-DP levels: >1000 femtomole per blood spot (fmol/punch). For participants taking emtricitabine/tenofovir alafenamide this will be TFV-DP levels: >140 femtomole per blood spot (fmol/punch).
Time Frame: 12-month follow up
Population: Participants with biomarker data indicating adherent daily PrEP dosing. For participants either reporting the use of both medications in the period or not reporting which medication they used during this time, investigators used decision rules to determine adherence. For instance, if a participant had a TFV-DP level above both cutpoints, they would be classified as adherent.
Measure: Count of Participants; unit: Participants
Arm/Group | ePrEP | Standard of Care
Number analyzed (Participants) | 37 | 48
Participants | 15 | 20

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time consent to participate in the study was given, during study participation up to 12 months.
Arm/Group | ePrEP | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/109
Other Adverse Events (participants affected / at risk) | 1/108 | 0/109
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ePrEP (N=108) | Standard of Care (N=109)
Increase in serum creatinine level (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03729570/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT03729570/ICF_001.pdf